CLINICAL TRIAL: NCT06398444
Title: A Clinical Study to Evaluate the Safety and Efficacy of Lutetium[177Lu] Oxodotreotide Injection in Patients With Advanced Somatostatin Receptor Positive Neuroendocrine Neoplasms
Brief Title: A Clinical Study of Lutetium[177Lu] Oxodotreotide Injection in Patients With Advanced Neuroendocrine Neoplasms
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XT-XTR008-2-02
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Advanced Neuroendocrine Neoplasm
MeSH Terms: interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lutetium[177Lu] Oxodotreotide Injection (Experimental)
  Interventions: Drug: Lutetium[177Lu] Oxodotreotide Injection

INTERVENTIONS:
Drug: Lutetium[177Lu] Oxodotreotide Injection — Participants will receive 7.4GBq (200mCi) Lutetium[177Lu] Oxodotreotide Injection every 8 weeks.

SUMMARY:
This is a multicenter, single-arm, two-part study designed to evaluate the safety and efficacy of Lutetium [177Lu] Oxyoctreotide Injection in patients with inoperable, locally advanced or metastatic, progressive, advanced somatostatin receptor (SSTR) positive neuroendocrine neoplasms (NEN) other than grade G1/G2 gastroenteropancreatic neuroendocrine tumors (GEP-NET).

DETAILED DESCRIPTION:
This study consists of two parts, the exploratory study (Part 1) and the pivotal study (Part 2).

In both parts, participants who signs Informed consent form (ICF) and is eligible for the study will be enrolled. Participants will receive 7.4GBq (200mCi) Lutetium [177Lu] Oxyoctreotide every 8 weeks. The objective tumor response will be assessed every 12 weeks from the time of the first dose according to RECIST 1.1 until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and have willingness to provide a written informed consent document.
2. Aged 18 years or older.
3. ECOG performance status 0 or 1.
4. Histopathologically confirmed, unresectable locally advanced or metastatic NEN .
5. Disease progression before first dose.
6. Subjects of childbearing potential should voluntarily use an effective method of contraception during treatment and within 4 months (male) or 7 months (female) of the last dose.

Exclusion Criteria:

1. Known brain metastases, unless these metastases have been treated and stabilized for at least 24 weeks prior to enrollment in the study.
2. Uncontrolled congestive heart failure, including baseline left ventricular ejection fraction (LVEF) <50%.
3. Uncontrolled diabetes mellitus, including baseline fasting glucose > 2 x ULN.
4. Any clinically significant active infection.
5. Pregnant or lactating females.
6. Received systemic antitumor therapy such as targeted therapy, immunotherapy, antitumor herbal therapy or chemotherapy within 4 weeks prior to enrollment.
7. Known other malignancies (except for those without recurrence within 5 years after adequate treatment).
8. Any other disease, mental status or surgical condition that is uncontrolled, may interfere with study completion (including poor compliance) or is inappropriate for the use of the investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AE) (Part1) | Until 6 months after the last dose
Overall Response Rate (ORR) assessed by Independent Review Committee (IRC) (Part 2) | Until disease progression or death, up to 5 years

SECONDARY OUTCOMES:
Overall Response Rate (ORR) (Part 1) | Until disease progression or death, up to 5 years
Progression-free survival (PFS) (Part 1) | Until disease progression or death, up to 5 years
Disease Control Rate (DCR) (Part 1) | Until disease progression or death, up to 5 years
Duration of Overall Response (DoR) (Part 1) | Until disease progression or death, up to 5 years
Time to Progression (TTP) (Part 1) | Until disease progression or death, up to 5 years
PFS rate at 12 months (Part 1) | At 12 months after the first dose
Overall Survival (OS) (Part 1) | Until death of any cause, up to 5 years
Change From Baseline in the EORTC QLQ-C30 Questionnaire (Part 1) | Until disease progression or death, up to 5 years
Change From Baseline in the EORTC Quality of Life Questionnaire (Part 1) | Until disease progression or death, up to 5 years
Progression-free survival (PFS) (Part 2) | Until disease progression or death, up to 5 years
Disease Control Rate (DCR) (Part 2) | Until disease progression or death, up to 5 years
Duration of Overall Response (DoR) (Part 2) | Until disease progression or death, up to 5 years
Time to Progression (TTP) (Part 2) | Until disease progression or death, up to 5 years
PFS rate at 12 months (Part 2) | At 12 months after the first dose
Overall Survival (OS) (Part 2) | Until death of any cause, up to 5 years
Change From Baseline in the EORTC QLQ-C30 Questionnaire (Part 2) | Until disease progression or death, up to 5 years
Change From Baseline in the EORTC Quality of Life Questionnaire (Part 2) | Until disease progression or death, up to 5 years
Incidence and severity of AE (Part2) | Until 6 months after the last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No